CLINICAL TRIAL: NCT05782023
Title: Supporto Alla Prevenzione Cardiovascolare Secondaria Post-IAM Attraverso un Programma di Empowerment Web-based (PREVEN-IAM)
Brief Title: Secondary Cardiovascular Prevention Post-acute Myocardial Infarction (AMI) Through a Web-based Empowerment Program
Acronym: PREVEN-IAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, José Pablo Werba, Principal Investigator, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCM 1547
Record Dates: First submitted 2023-02-21; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; secondary prevention; atherosclerosis; health empowerment
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital empowerment (Experimental): Usual-care + preventive intervention through digital empowerment
  Interventions: Behavioral: Digital empowerment
- Usual care (No Intervention): Usual-care (cardiologist visit at 1, 3 and 12 months after AMI)

INTERVENTIONS:
Behavioral: Digital empowerment — The intervention will consist of a minimal interaction face-to-face before hospital discharge for risk factors profiling followed by actions for health empowerment, delivered through an ad-hoc developed web platform, which include: a) periodic delivery of email messages with links to educational, motivational and supportive materials for secondary prevention, b) access to a message box for questions and answers and c) possibility of video-calls with the preventive team.
  Arms: Digital empowerment

SUMMARY:
The aim of this study is to assess the efficacy of an innovative program of secondary cardiovascular prevention focused on patient empowerment. This program will be characterized by a blended interaction between healthcare workers and the patients: first, a face-to-face first encounter in-hospital for risk factors profiling, followed by remote interactions through a digital approach. The digital intervention is targeted at promoting the adoption and retention of virtuous behavior (e.g. smoking cessation, healthy eating habits, physical exercise, regular assumption of pharmacological therapies), improving cardiovascular risk factors control. Moreover, an exploratory endpoint will be investigated: the reduction of the residual coronary risk.

DETAILED DESCRIPTION:
The experimental intervention will consist of educational, motivational and coaching actions of patients post-AMI through a web based interaction with the prevention team. This intervention will be: 1) personalized (based on a risk factor profile obtained in-hospital) 2) agreed (planned with the patient with shared decision making), 3) multidisciplinary (physician, nutritionist, psychologist, clinical research nurse), 4) blended, composed of a minimal initial interaction face-to-face and periodical reminders (educational, motivational and supportive) for secondary prevention, through email, a reserved website and a chat box. The intervention contents, targeted at patient empowerment, will take the behavioral change models into consideration as a theoretical basis.

The participants of both groups will undergo conventional cardiology follow-up visits indicated (at 1- 3-12-36-48 months). Blood tests or any other exam other than those indicated by routine clinical practice are not required in this study. Patients with diabetes who already wear the Abbot Freestyle Libre® glucose monitoring device will be asked access to device data within two periods of two weeks, before programmed cardiology visits at 1, 3 and 12 months. At 12 months and 48 months-follow-up visits, all participants will be assessed by the Atherosclerosis Prevention Unit, and the lifestyle questionnaires administered at baseline will be repeated. The intervention group will also take a satisfaction survey at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* STEMI or NSTEMI
* availability of digital communication devices (smart-phone, tablet or personal computer) and internet access

Exclusion Criteria:

* active malignancies (except for skin tumors other than melanoma)
* life expectancy <5 years
* absolute clinical indication to undergo hospital rehabilitation cycles
* cognitive status undermining digital communication devices use, even after proper training
* low understanding of Italian language, either oral or written, by clinician's judgement
* patient not foreseeing to undergo cardiology follow-up at the site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy on measurable risk factors - BMI | 12 months
  Measured through the changes in the BMI, measured in weight in kilograms divided by the square of height in meters (kg/m2).
Efficacy on measurable risk factors - systolic blood pressure | 12 months
  Measured through the changes in the systolic blood pressure, measured in millimetres (mm) of mercury (Hg) (mmHg).
Efficacy on measurable risk factors - diastolic blood pressure | 12 months
  Measured through the changes in the diastolic blood pressure, measured in millimetres (mm) of mercury (Hg) (mmHg).
Efficacy on measurable risk factors - LDL-cholesterol levels | 12 months
  Measured through the changes in the LDL-cholesterol levels, measured in milligrams per deciliter (mg/dL).
Efficacy on measurable risk factors - glycemia levels | 12 months
  Measured through the changes in the glycemia levels, measured in milligrams per deciliter (mg/dL).
Efficacy on measurable risk factors - glycosylated hemoglobin in diabetic patients | 12 months
  Measured through the changes in the glycosylated hemoglobin in diabetic patients, measured in percentage (%) of glycosylated hemoglobin over total hemoglobin, or in millimole of glycated hemoglobin per mole of total hemoglobin (mmol/mol).
Efficacy on measurable risk factors - expired carbon monoxide in smokers | 12 months
  Measured through the changes in the expired carbon monoxide (CO) in smokers, measured in parts of expired carbon monoxide per million (ppm) per hour (ppm/h), assessed through the Smokerlyzer®.

SECONDARY OUTCOMES:
Efficacy on lifestyle changes - physical activity | 12 months
  Measured through the International Physical Activity Questionnaires (IPAQ). Based on the responses, three categories are identified:
  1. Inactive
     * No activity is reported OR
     * Some activity is reported but not enough to meet categories 2 or 3.
  2. Minimally Active
     Any one of the following 3 criteria:
     * ≥3 days of vigorous activity of ≥20 minutes per day OR
     * ≥5 days of moderate-intensity activity or walking of ≥30 minutes per day OR
     * ≥5 days of any combination of walking, moderate-intensity or vigorous intensity activities achieving ≥600 MET-min/week.
  3. HEPA (health enhancing physical activity) active
  Anyone of the following 2 criteria:
  * Vigorous-intensity activity on ≥3 days and accumulating ≥1500 METminutes/week OR
  * ≥7 days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum of ≥3000 MET-minutes/week.
Efficacy on lifestyle changes - adherence to a "heart-friendly" diet | 12 months
  Measured through the Mediterranean Diet Adherence Screener (MEDAS). The final MEDAS score can range between 0 and 14. To categorize the overall MEDAS score, a cut-off score of ≥8 points is used to denote adherence to the principles of the mediterranean diet, while MEDAS score of ≤7 points represents mediterranean diet non-adherence.
Efficacy on lifestyle changes - smoking reduction or cessation | 12 months
  Measured through the number of smoked cigarettes.
Efficacy on lifestyle changes - self-efficacy | 12 months
  Measured through the General Self-Efficacy Scale, GSE. It is composed of 10 items, and the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Efficacy on lifestyle changes - Health Locus of Control | 12 months
  Measured through the Multidimensional Health Locus of Control (MHLC) questionnaire. The survey has 18 items with 6 items for each of its 3 subscales: Internal, Chance and Powerful Others. Each item is scored on a 6 point, Likert-type scale.
  The Internal subscale measures the strength of the belief that the respondent's health is the result of their own behaviors: higher scores indicate a more Internal Health Locus of Control, lower scores indicate a more External Health Locus of Control.
  The Powerful Others subscale measures the degree to which the respondent believes health is controlled by clinicians or a higher power. The Chance subscale indicates the degree to which the respondent believes that health is out of their control. Higher scores on both the Powerful Others and Chance subscales represent a more External Health Locus of Control while lower scores on the Powerful Others and Chance subscales indicate a more Internal Health Locus of Control.
Efficacy on cardioprotective treatment adherence | 12 months
  Measured through the Morisky Medication Adherence Scale (MMAS-8). The MMAS-8 range from 0 to 8, with scores of 8 reflecting high adherence, 7 or 6 reflecting medium adherence, and <6 reflecting low adherence.
Efficacy on glucose control in diabetic patients | 12 months
  Measured in diabetic patients who already use the continuous monitoring device Abbott Freestyle Libre® as the variation of the following parameters, to be considered 2 weeks before and after the educational intervention:
  * mean glycemia (mg/dl)
  * Glucose Management Indicator (GMI) (mmol/mol or %)
  * glycemic variability (measured through the glycemic variability coefficient during monitoring, %)
  * Time In Range (TIR) (70-180 mg/dl)
  * High Time In Range (HTR) (>180 mg/dl)
  * Low Time In Range (LTR) (<70 mg/dl)
  * hyperglycemia or hypoglycemia episodes ≥15 min within the area under the curve
Long-term maintenance of controlled levels of risk factors - BMI | 48 months
  Measured through the changes in the BMI, measured in weight in kilograms divided by the square of height in meters (kg/m2).
Long-term maintenance of controlled levels of risk factors - systolic blood pressure | 48 months
  Measured through the changes in the systolic blood pressure, measured in millimetres (mm) of mercury (Hg) (mmHg).
Long-term maintenance of controlled levels of risk factors - diastolic blood pressure | 48 months
  Measured through the changes in the diastolic blood pressure, measured in millimetres (mm) of mercury (Hg) (mmHg).
Long-term maintenance of controlled levels of risk factors - LDL cholesterol | 48 months
  Measured through the changes in the LDL-cholesterol levels, measured in milligrams per deciliter (mg/dL).
Long-term maintenance of controlled levels of risk factors - glycemia levels | 48 months
  Measured through the changes in the glycemia levels, measured in milligrams per deciliter (mg/dL).
Long-term maintenance of controlled levels of risk factors - glycosylated hemoglobin in diabetic patients | 48 months
  Measured through the changes in the glycosylated hemoglobin in diabetic patients, measured in percentage (%) of glycosylated hemoglobin over total hemoglobin, or in millimole of glycated hemoglobin per mole of total hemoglobin (mmol/mol).
Long-term maintenance of controlled levels of risk factors - expired carbon monoxide in smokers | 48 months
  Measured through the changes in the expired carbon monoxide (CO) in smokers, measured in parts of expired carbon monoxide per million (ppm) per hour (ppm/h), assessed through the Smokerlyzer®.
Efficacy on secondary prevention | 48 months
  Measured as the incidence of symptomatic coronary events (exploratory analysis).

CONTACTS AND LOCATIONS:
Overall Officials: José P Werba, MD, Principal Investigator — Centro Cardiologico Monzino
Locations (1):
- Centro Cardiologico Monzino, Milan, Italy